CLINICAL TRIAL: NCT01553435
Title: Effect of N-methyl D-aspartate (NMDA) Receptor Antagonist Dextromethorphan on Opiods Analgesia and Tolerance in Pediatric Intensive Care Unit Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Principal Investigator, Mohammed Naeem, Consultant Pediatric Intensivist, King Abdullah International Medical Research Center
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: RC 09-120
Record Dates: First submitted 2012-03-06; First posted 2012-03-14 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Pain; Opioid Tolerance; Analgesia Tolerance
Keywords: Dextromethorphan; Morphine; Fentanyl; Opioid; analgesia; Efficacy
MeSH Terms: conditions — Pain; Agnosia | interventions — Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dextromethorphan, opioid analgisia, efficacy (Placebo Comparator)
  Interventions: Drug: Dextromethorphan
- Placebo,opioid analgesia, efficacy (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dextromethorphan — The study medicines shall be administered via tube.
  Arms: Dextromethorphan, opioid analgisia, efficacy
Drug: Placebo — The study medicines shall be administered via tube.
  Arms: Placebo,opioid analgesia, efficacy

SUMMARY:
Effect of N-methyl D-aspartate (NMDA) receptor antagonist Dextromethorphan on Opiods analgesia and tolerance in Pediatric Intensive Care Unit Patients

ELIGIBILITY:
Inclusion:

* Patients above 2 years, admitted in PICU
* On Morphine or Fentanyl infusions for more than 48 hours

Exclusion Criteria:

* Patients under 2 years of age
* Patients with anticipated PICU length of stay less than 3 days.
* Patients shall be excluded if Morphine or Fentanyl infusions not continued for the minimum duration of 72 hours after enrollment
* Patients develops hemodynamic instability
* Patients with Hepatic failure
* Withdrawal request by parent(s)/guardian/family

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2011-01; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Effect of N-methyl D-aspartate (NMDA) receptor antagonist Dextromethorphan on Opiods analgesia and tolerance in Pediatric Intensive Care Unit Patients | Two years
  Control of pain

SECONDARY OUTCOMES:
Effect of N-methyl D-aspartate (NMDA) receptor antagonist Dextromethorphan on Opiods analgesia and tolerance in Pediatric Intensive Care Unit Patients | two years
  Duration of ventilation in both groups
Effect of N-methyl D-aspartate (NMDA) receptor antagonist Dextromethorphan on Opiods analgesia and tolerance in Pediatric Intensive Care Unit Patients | Two years
  Length of Hospital Stay in two groups

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdul Aziz Medical City, Riyadh, Central, Saudi Arabia

REFERENCES:
- [Derived] Naeem M, Al Alem H, Al Shehri A, Al-Jeraisy M. Effect of N-Methyl-D-Aspartate Receptor Antagonist Dextromethorphan on Opioid Analgesia in Pediatric Intensive Care Unit. Pain Res Manag. 2016;2016:1658172. doi: 10.1155/2016/1658172. Epub 2016 Oct 27. PMID 27867308